CLINICAL TRIAL: NCT03718949
Title: Can Continuous Cardiac Output Monitoring Before General Anesthesia Predict Hypotension After Induction?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201807139DIPB
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-10

CONDITIONS: Anesthesia, General; Hypotension; Cardiac Output
Keywords: pre-operative fasting; general anesthesia; cardiac output,Ultrasonography; Ultrasonography
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Post-induction hypotension (PIH) is very common with high incidence about 9-60%. There are multiple factors that may cause PIH, like pre-operative fasting, bowel preparation, vasodilatation due to anesthetics, and reduced stimulation during preparation before incision. Hypotension could cause tissue hypoperfusion, ischemia and higher risk for stroke or myocardial infarction, which result in higher risk for prolonged hospital stay or death. In general surgical patients, lower pre-induction SAP, older age (>50 years old), and emergency surgery are independently associated with PIH. In this study, we would like to use a wireless continuous non-invasive sonography device to evaluate if the change of cardiac output during the perioperative period could predict PIH.

Ｗe would like to enroll 80 patients of ASA class I to III who undergo abdominal surgery. GIS-Heartio® will be used to estimate the cardiac parameters one day before the surgery (Day 0) and after the patient enter the operation room till wound incision. Passive leg raise test would be performed on day 0 and before induction. We will analyze the patient's demographic data and the cardiac parameters to see if continuous cardiac output monitor can predict the occurrence of PIH.

DETAILED DESCRIPTION:
Post-induction hypotension (PIH) is very common with high incidence about 9-60% in every kind of surgeries includes general anesthesia and neuraxial anesthesia. There are multiple factors that may cause PIH, like pre-operative fasting, bowel preparation, vasodilatation due to anesthetics, sympathetic blockade and reduced stimulation during preparation before surgical incision. Hypotension during the surgeries could possibly cause tissue hypoperfusion, tissue ischemia and higher risk for acute kidney failure, stroke or myocardial infarction, which result in higher risk for prolonged hospital stay or death [1-4]. In general surgical patients, lower pre-induction systolic arterial pressure, older age (>50 years old), and emergent surgery are independently associated with PIH[1].

However, nowadays heart rate variability (HRV), the inferior vena cava(IVC) ultrasound, and stroke volume variation were demonstrated to be able to predict the PIH event [5-7]. However, people with any kind of arrhythmia is not suitable for HRV analysis. Part of obese patients are not suitable for IVC ultrasound due to poor image quality. Stroke volume variation can only be monitored if the arterial catheter and Flotrac® were applied on the patient before anesthetic induction.

In this study, the wireless continuous non-invasive sonography device has the benefits of light-weighted, short learning curve, non-invasive, continuous monitoring, and more intuitive collected data. It's a huge progress for non-invasive cardiac output during anesthesia with GIS-Heartio®. The primary endpoint is if the change of cardiac output after fasting could predict PIH. The second endpoint is whether the change of cardiac output during "passive leg test" could predict PIH. If PIH can be predicted and prevented before anesthesia, the safety of the surgery and prognosis of patient will be elevated!

ELIGIBILITY:
1. >20 years old
2. American Society of Anesthesiologists Classification(ASA) I~III
3. patients accept major surgery under general anesthesia, and monitored with invasive arterial blood pressure and estimated cardiac output.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients older than 20 years old, and accept major surgery
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-12-04 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
post-induction hypotension | 20 minutes after induction
  mean arterial blood pressure 30% lower than baseline, or mean arterial blood pressure <60mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Tzu Li, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan